CLINICAL TRIAL: NCT01335165
Title: A Phase 1, Single Ascending Dose Study of the Safety and Pharmacokinetics of TT30 in Subjects With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Brief Title: Safety and Pharmacokinetics of TT30 in Subjects With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inability to reach enrollment as planned
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TT30-PNH-002
Record Dates: First submitted 2011-04-12; First posted 2011-04-14 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
Keywords: PNH
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TT30 (ALXN1102 Formulation) (Experimental): IV: 0.1, 0.3, and 1.0 mg/kg
  Interventions: Drug: ALXN1102
- TT30 (ALXN1103 Formulation) (Experimental): IV: 3.0, 6.0, and 10.0 mg/kg
  SC: 1.0 and 3.0 mg/kg
  Interventions: Drug: ALXN1103

INTERVENTIONS:
Drug: ALXN1102 — Single Ascending Dose IV
  Arms: TT30 (ALXN1102 Formulation)
Drug: ALXN1103 — Single Ascending Dose IV or SC
  Arms: TT30 (ALXN1103 Formulation)

SUMMARY:
The purpose of this research study is to understand the safety, pharmacokinetics and pharmacodynamics of a single dose of TT30 (ALXN1102 and ALXN1103 formulations) when given IV (through a vein) or SC (under the skin) to patients with PNH.

DETAILED DESCRIPTION:
This is an open-label, single-dose, dose-escalation study to assess the safety, tolerability, PK, PD, and immunogenicity of TT30 given as an IV infusion and as a SC injection in subjects with PNH or evidence of circulating PNH cells.

Eligible subjects with PNH will be vaccinated with meningococcal vaccine at least two weeks prior to dosing (if not previously vaccinated or if revaccination is required).

On study day 1, the subject will receive the single dose of TT30 as an IV infusion over 60 minutes or as a SC injection, and be followed with additional study evaluations over the next 59 days.

ELIGIBILITY:
Inclusion Criteria:

* Individuals at least 18 years of age with a diagnosis of PNH & vaccination against meningococcus.

Exclusion Criteria:

* Abnormal renal or liver function
* History of meningococcal disease
* History of Guillain-Barre syndrome
* Known infection with HIV or Hepatitis B or C
* History of thrombotic events

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Assess the safety and tolerability of a single dose of TT30. | 60 days
  Safety and tolerability will be evaluated in all subjects by physical exam, vital signs, ECGs, laboratory changes over time, adverse events, and antibody development.

SECONDARY OUTCOMES:
Characterize PK, PD and immunogenicity of a single dose of TT30. | 60 days
  Immunogenicity will be will be assessed using standard measures for these parameters. PK and PD will be assessed by using standard measures, including reticulocyte count and lactate dehydrogenase (LDH) levels.

CONTACTS AND LOCATIONS:
Overall Officials: Bill Lundberg, MD, Study Director — Alexion Pharmaceuticals, Inc.
Locations (5):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States
- Institute of Hematology and Blood Transfusion / Institut Hematologie a krevní transfuze, U Nemocnice 1, Prague 2, Czechia
- Federico II University of Naples, Via Pansini 5, Naples, Italy
- University Clinical Centre, Dębinki, Gdańsk, Poland
- King's College Hospital NHS Foundation Trust, Denmark Hill, London, United Kingdom